CLINICAL TRIAL: NCT00059995
Title: Phase I/II Open Label, Dose-Escalating Study of MDX-060 Administered Weekly for 4 Weeks in Patients With Refractory/Relapsed CD30 Lymphoma
Brief Title: MDX-060 Monoclonal Antibody in Treating Patients With Refractory or Relapsed Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: MDX-060-01; MSKCC-02121; CDR0000298995 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2009-11

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; anaplastic large cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent childhood large cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Recurrence; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Large B-Cell, Diffuse; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous | interventions — iratumumab

INTERVENTIONS:
Biological: iratumumab

SUMMARY:
RATIONALE: Monoclonal antibodies such as MDX-060 can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

PURPOSE: Phase I/II trial to study the effectiveness of MDX-060 monoclonal antibody in treating patients who have refractory or relapsed lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of MDX-060 monoclonal antibody in patients with refractory or relapsed CD30-positive lymphoma.
* Determine the maximum tolerated dose and dose-limiting toxicity of this drug in these patients.
* Determine the pharmacokinetic profile of this drug in these patients.
* Determine, preliminarily, the efficacy (antilymphoma activity) of this drug in these patients.

OUTLINE: This is an open-label, multicenter, dose-escalation study.

Patients receive MDX-060 monoclonal antibody IV over 90 minutes once weekly for 4 weeks.

Cohorts of 3-6 patients receive escalating doses of MDX-060 monoclonal antibody until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional 16 patients are accrued and receive MDX-060 monoclonal antibody at the MTD.

Patients are followed monthly for 3 months and then every 3 months for 18 months or until disease progression.

PROJECTED ACCRUAL: A maximum of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed B-cell or T-cell lymphoma

  * Hodgkin's lymphoma and anaplastic large cell lymphoma eligible
  * No HIV-associated lymphoma
* CD30-positive disease by biopsy, flow cytometry, or immunohistochemistry

  * At least 50% of malignant cells (specifically Reed-Sternberg cells for Hodgkin's lymphoma) must express CD30
* Must meet one of the following criteria for relapsed/refractory disease:

  * Relapsed after prior chemotherapy or radiotherapy and autologous or allogeneic bone marrow transplantation (if appropriate)

    * Relapsed disease must be within the prior irradiated field
  * Disease that is refractory to prior chemotherapy or radiotherapy with no other curative treatment option

    * Disease progression must be within the prior irradiated field
* Progressive and evaluable disease (measurable disease required for patients accrued on study after the maximum tolerated dose is determined)

PATIENT CHARACTERISTICS:

Age

* Over 12

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* WBC at least 1,500/mm^3*
* Neutrophil count at least 1,000/mm^3*
* Platelet count at least 75,000/mm^3*
* Hemoglobin at least 8.0 g/dL* NOTE: *Laboratory abnormalities attributable to organ involvement by lymphoma are allowed

Hepatic

* AST no greater than 2 times upper limit of normal (ULN)*
* Bilirubin no greater than 2.0 mg/dL (unless due to Gilbert's syndrome)*
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative NOTE: *Laboratory abnormalities attributable to organ involvement by lymphoma are allowed

Renal

* Creatinine no greater than 2 times ULN* NOTE: *Laboratory abnormalities attributable to organ involvement by lymphoma are allowed

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 9 months after study participation
* HIV negative
* No other active malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No active significant infection
* No apparent opportunistic infection, as indicated by any of the following:

  * Purified protein derivative recently determined to be positive
  * Infectious infiltrate by chest x-ray
  * Recent changes in fever/chill patterns
  * New, unexplained neurological symptoms
* No underlying medical condition that would preclude receiving study therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior anti-CD30 antibody therapy
* No other concurrent biologic therapy

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* No concurrent systemic steroidal therapy (excluding physiologic doses)

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* Not specified

Other

* No other concurrent investigational agents

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-01; Primary Completion 2007-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Horwitz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio

REFERENCES:
- [Result] Ansell SM, Horwitz SM, Engert A, Khan KD, Lin T, Strair R, Keler T, Graziano R, Blanset D, Yellin M, Fischkoff S, Assad A, Borchmann P. Phase I/II study of an anti-CD30 monoclonal antibody (MDX-060) in Hodgkin's lymphoma and anaplastic large-cell lymphoma. J Clin Oncol. 2007 Jul 1;25(19):2764-9. doi: 10.1200/JCO.2006.07.8972. Epub 2007 May 21. PMID 17515574